CLINICAL TRIAL: NCT06757010
Title: A Double-Blind, Randomized, Placebo-controlled, Study of NE3107 in Subjects With Early Parkinson's Disease
Brief Title: A Study of NE3107 in Early Parkinson's
Acronym: SUNRISE-PD
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: BioVie Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NE3107-PD-202
Record Dates: First submitted 2024-12-24; First posted 2025-01-03 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Parkinsons Disease (PD)
Keywords: Treatment naïve Parkinson's; Early Parkinson's
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- NE3107 (Experimental): Subjects will receive 20 mg NE3107 BID (twice daily administration; 40 mg daily) as oral capsules.
  Interventions: Drug: NE3107
- Placebo (Placebo Comparator): Subjects will receive matching placebo capsules for oral administration BID (twice daily).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: NE3107 — NE3107 20 mg BID
  Other Names: bezisterim
  Arms: NE3107
Drug: Placebo — Placebo BID
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to learn if bezisterim can treat movement symptoms of Parkinson's disease in patients that are 45 to 80 years old, in generally good physical and mental health, and are nearing the need for treatment to relieve their symptoms but have not yet been prescribed any form of levodopa or drug with similar activity. The main questions it aims to answer are:

* Will bezisterim decrease movement symptoms of Parkinson's disease?
* What medical problems do participants have when taking bezisterim?

Researchers will compare the effects of bezisterim treatment to placebo (a look-alike substance that contains no drug) to see if bezisterim works to treat movement symptoms of Parkinson's disease.

Participants will

* have a physical examination that includes an electrocardiogram
* take drug or placebo twice daily for four months
* visit a clinical site or receive an at home visit seven times over the course of five months

ELIGIBILITY:
Inclusion Criteria:

* 45 years to 80 years of age
* diagnosed with idiopathic Parkinson's Disease (PD) within 18 months
* nearing the need for symptomatic therapy
* agree to use birth control measures
* provide voluntary consent
* willing to allow blood collection for DNA methylation analysis
* pass all screening tests and procedures

Exclusion Criteria:

* has taken levodopa or another similar drug for the motor symptoms of PD
* a known or strongly suspected familial cause for PD diagnosis
* major mental health or physical illness
* medical history of major mental or physical illness

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-03-26 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-01-02 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in the MDS-UPDRS Part III | 12 Weeks
  The Movement Disorder Society-Unified Parkinson's Disease Rating Scale (MDS-UPDRS) is comprised of 4 parts: This study will use MDS-UPDRS Parts I, II, and III. The primary efficacy endpoint is change in the modified MDS-UPDRS Part III score. Scores (0-4: Normal to severe impact) are derived from clinician and subject input to allow the assessment of symptomatic worsening, stability, or improvement.

SECONDARY OUTCOMES:
Change from baseline in MDS-UPDRS Part I and II | 12 weeks
  The Movement Disorder Society-Unified Parkinson's Disease Rating Scale (MDS-UPDRS) is comprised of 4 parts: This study will use MDS-UPDRS Parts I, II, and III.
  Secondary efficacy endpoints in the study will include change in the modified MDS-UPDRS Part I and II scores. Scores (0-4: Normal to severe impact) are derived from clinician and subject input to allow the assessment of symptomatic worsening, stability, or improvement.
Percent of subjects with improvement in Clinical Global Impression | 12 weeks
  Percent of subjects with any improvement as measured by Clinical Global Impression.

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Quest Research Institute, Farmington Hills, Michigan
  - Dent Neurologic, Amherst, New York
  - Science 37 (Nationwide Site), Morrisville, North Carolina
  - NeuroScience Research Center, LLC, Canton, Ohio

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: www.SunrisePD.com — https://sunrisepd.com/